CLINICAL TRIAL: NCT01006226
Title: A Pilot Study of 64CuATSM and Hypoxia in Stage IV Non-small Cell Lung Cancer Patients Treated With Carboplatin, Paclitaxel, and Bevacizumab
Brief Title: 64CuATSM and Hypoxia in Stage IV Non-small Cell Lung Cancer With Carboplatin, Paclitaxel, and Bevacizumab
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to funding issues
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-1640
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 64Cu-ATSM PET (Experimental)
  Interventions: Drug: 64Cu-ATSM PET

INTERVENTIONS:
Drug: 64Cu-ATSM PET — 2 64Cu-ATSM PET scan, one pretreatment and one 19-21 days after the first dose of bevacizumab

SUMMARY:
The purpose of this study is to determine:

* Whether bevacizumab increases the amount of oxygen in cancer as measured by a special positron emission tomography (PET) scan using 64Cu-ATSM.
* Whether the amount of oxygen in cancer as measured by 64Cu-ATSM PET scan predicts how well the cancer responds to treatment with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-squamous NSCLC.
* Clinically or pathologically proven Stage IV NSCLC.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm irrespective of scanner type.
* No previous chemotherapy.
* Age >18 years.

Because no dosing or adverse event data are currently available on the use of 64Cu-ATSM in combination with paclitaxel, carboplatin, and bevacizumab in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric phase 2 combination trials.

* ECOG performance status 0-1.
* Patients must have normal organ and marrow function as defined below:
* hemoglobin >9 gm/dL
* absolute neutrophil count >1,500/mcL
* platelets >100,000/mcL
* total bilirubin < 1.5 mg/dL
* AST(SGOT)/ALT(SGPT) <3 X institutional upper limit of normal
* alkaline phosphatase <3 X institutional upper limit of normal
* creatinine <1.5 X institutional upper limit of normal

OR

* creatinine clearance >60 mL/min/1.73 m2 (Cockcroft Gault)
* urine dipstick for proteinuria < 1+
* Adequate coagulation function - INR < 1.5 and PTT < institutional upper limit of normal.
* The effects of 64Cu-ATSM on the developing human fetus at the recommended imaging dose are unknown. For this reason and because chemotherapeutic agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability of the patient to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had prior chemotherapy.
* Patients who have had prior radiation therapy for lung cancer.
* Patients may not be receiving any other investigational agents.
* Patients with known central nervous system metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 64Cu-ATSM or other agents used in the study.
* History of claustrophobia, since patients might not be able to tolerate 64CuATSM-PET imaging.
* History of gross hemoptysis - bright red blood of > ½ teaspoon in quantity - in past 6 months.
* Any concurrent or history of active malignancy in the prior five years except for basal cell skin cancer or carcinoma in situ of the cervix.
* History of thrombotic or hemorrhagic disorder.
* Anticoagulation at treatment/therapeutic doses.
* Uncontrolled hypertension.
* Pre-existing neuropathy > grade 1.
* Treatment with aspirin > 325 mg/day, dipyridamole, ticlopidine, clopidogrel, and/or cilostazol that cannot be discontinued.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because paclitaxel, carboplatin, and bevacizumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with paclitaxel, carboplatin, and bevacizumab, breastfeeding should be discontinued if the mother is treated with these agents. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To determine whether bevacizumab improves tumor hypoxia as measured by 64Cu-ATSM-PET in patients with previously untreated metastatic NSCLC. | 3 years

SECONDARY OUTCOMES:
To determine whether bevacizumab and chemotherapy improves response rates in tumors defined to be hypoxia by 64-Cu-ATSM-PET in patients with treatment-naïve NSCLC than what would be expected with chemotherapy alone. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria Baggstrom, M.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu